CLINICAL TRIAL: NCT00276601
Title: A Pilot Study of Arsenic Trioxide-Based Consolidation Therapy for the Primary Treatment of Acute Promyelocytic Leukemia
Brief Title: Combination Chemotherapy in Treating Patients With Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven D. Gore, Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Purpose: Treatment
Other Study IDs: J0442, CDR0000449985; P30CA006973 (NIH); JHOC-J0442; WIRB-20041058
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Cytarabine; Daunorubicin; Mercaptopurine; Methotrexate; Tretinoin

INTERVENTIONS:
Drug: arsenic trioxide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy works in treating patients with acute promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, preliminarily, the safety of incorporating arsenic trioxide (ATO) into cytarabine and daunorubicin hydrochloride-based consolidation therapy followed by tretinoin maintenance therapy in patients receiving induction tretinoin and daunorubicin hydrochloride with acute promyelocytic leukemia (APL) induced into remission with tretinoin and daunorubicin hydrochloride.
* Determine, preliminarily, the efficacy of this strategy in inducing and maintaining molecular remissions in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

* Induction therapy: Patients receive oral tretinoin twice daily on days 1-60 and daunorubicin hydrochloride IV on days 4, 6, and 8. Patients are evaluated between days 60-67 and proceed to consolidation therapy.
* Consolidation therapy: Patients receive cytarabine IV continuously on days 1-3, daunorubicin hydrochloride IV on days 1-3, and arsenic trioxide IV over 1-2 hours once daily, 5 days a week, beginning on day 8 and continuing for 6 weeks. Patients with clinical and/or cytogenic, but not molecular, remission receive additional arsenic trioxide once daily, 5 days a week, for 30 doses (6 weeks). Patients achieving clinical and molecular remission after completion of 6 or 12 weeks of arsenic trioxide proceed to maintenance therapy.
* Maintenance therapy: Patients receive oral tretinoin once daily on days 1-15. Treatment repeats every 3 months for 8 courses (2 years).

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute promyelocytic leukemia (APL) by morphologic and flow cytometric documentation (high orthogonal light scatter, lack of HLA-DR expression)

  * Patients with classical APL as well as the microgranular variant (M3V) are eligible

    * In cases where the diagnosis is unclear, consultation with a hematopathologist is required before enrolling the patient in the study
* Patients found to have cytogenetic abnormalities that do not produce the PML-RARα gene rearrangement will be removed from study and will not be included in data analysis

PATIENT CHARACTERISTICS:

* Patients will not be excluded because of performance status or comorbid disease
* Premenopausal female patients must have a negative pregnancy test

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for APL except hydroxyurea

Ages: 5 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 2 and 5 years after study completion
Safety of arsenic trioxide following cytarabine and anthracycline immediately after study completion

SECONDARY OUTCOMES:
Validate peripheral blood real-time PCR for minimal disease monitoring as measured by real-time PCR for PML-RARalpha monthly for two years after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Gore, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (7):
- United States (7):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania